CLINICAL TRIAL: NCT00912041
Title: BrainGate2: Feasibility Study of an Intracortical Neural Interface System for Persons With Tetraplegia
Acronym: BrainGate2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh R. Hochberg, MD, PhD. (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Leigh R. Hochberg, MD, PhD., Sponsor-Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MGH-BG2-TP-001; R01DC009899 (NIH); UH2NS095548 (NIH); A2295-R (Other Grant/Funding Number: U.S. Department of Veterans Affairs); U01NS123101 (NIH); R01DC014034 (NIH); U01DC017844 (NIH); CDMRP-AL220043 (Other Grant/Funding Number: Department of Defense (DOD)); A4820-R (Other Grant/Funding Number: U.S. Department of Veterans Affairs)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Tetraplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked in Syndrome; Muscular Dystrophy
Keywords: Brain computer interface; Assistive device; Environmental control; Communication device; quadriplegia; tetraplegia
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Locked-In Syndrome; Muscular Dystrophies | interventions — Neural Prostheses; Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- BrainGate (Other): BrainGate Neural Interface System
  Interventions: Device: Placement of the BrainGate2 sensor(s) into the motor-related cortex

INTERVENTIONS:
Device: Placement of the BrainGate2 sensor(s) into the motor-related cortex — Up to six 4x4 mm BrainGate2 sensor(s) are placed into the motor-related cortex (including speech-related areas of cortex), connected to one, two, or three percutaneous pedestals. Neural recordings are made at least weekly for a year or more.
  Other Names: BrainGate; NeuroPort; neural prosthesis; neural prosthetic; neuroprosthetic; brain computer interface; brain-computer interface

SUMMARY:
The purpose of this study is to obtain preliminary device safety information and demonstrate proof of principle (feasibility) of the ability of people with tetraplegia to control a computer cursor and other assistive devices with their thoughts.

DETAILED DESCRIPTION:
The goal of the BrainGate2 research and development project is to identify the core methods and features for a medical device that could allow people with paralysis, including severe speech impairment, to recover a host of abilities that normally rely on the hands or on speech.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinal cord injury, brainstem stroke, muscular dystrophy, amyotrophic lateral sclerosis or other motor neuron disorders
* Complete or incomplete tetraplegia (quadriplegia)
* Must live within a three-hour drive of the Study site
* (There are additional inclusion criteria)

Exclusion Criteria:

* Visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses
* Chronic oral or intravenous steroids or immunosuppressive therapy
* Other serious disease or disorder that could seriously affect ability to participate in the study
* (There are additional exclusion criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2009-05; Primary Completion 2038-09 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this Study is to determine the safety of the BrainGate2 Neural Interface System. | One year post-implant evaluation period

SECONDARY OUTCOMES:
To investigate the feasibility of BrainGate2 and to establish the parameters for a larger clinical study, such as appropriate neural decoding algorithms, sample size, indices of measurement, success criteria, and endpoints. | Course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Leigh R Hochberg, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - University of California, Davis, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Providence VA Medical Center, Providence, Rhode Island

REFERENCES:
- [Background] Hochberg LR, Serruya MD, Friehs GM, Mukand JA, Saleh M, Caplan AH, Branner A, Chen D, Penn RD, Donoghue JP. Neuronal ensemble control of prosthetic devices by a human with tetraplegia. Nature. 2006 Jul 13;442(7099):164-71. doi: 10.1038/nature04970. PMID 16838014
- [Background] Donoghue JP, Nurmikko A, Black M, Hochberg LR. Assistive technology and robotic control using motor cortex ensemble-based neural interface systems in humans with tetraplegia. J Physiol. 2007 Mar 15;579(Pt 3):603-11. doi: 10.1113/jphysiol.2006.127209. Epub 2007 Feb 1. PMID 17272345
- [Background] Homer ML, Perge JA, Black MJ, Harrison MT, Cash SS, Hochberg LR. Adaptive offset correction for intracortical brain-computer interfaces. IEEE Trans Neural Syst Rehabil Eng. 2014 Mar;22(2):239-48. doi: 10.1109/TNSRE.2013.2287768. PMID 24196868
- [Background] Perge JA, Zhang S, Malik WQ, Homer ML, Cash S, Friehs G, Eskandar EN, Donoghue JP, Hochberg LR. Reliability of directional information in unsorted spikes and local field potentials recorded in human motor cortex. J Neural Eng. 2014 Aug;11(4):046007. doi: 10.1088/1741-2560/11/4/046007. Epub 2014 Jun 12. PMID 24921388
- [Background] Masse NY, Jarosiewicz B, Simeral JD, Bacher D, Stavisky SD, Cash SS, Oakley EM, Berhanu E, Eskandar E, Friehs G, Hochberg LR, Donoghue JP. Non-causal spike filtering improves decoding of movement intention for intracortical BCIs. J Neurosci Methods. 2014 Oct 30;236:58-67. doi: 10.1016/j.jneumeth.2014.08.004. Epub 2014 Aug 13. PMID 25128256
- [Background] Malik WQ, Hochberg LR, Donoghue JP, Brown EN. Modulation depth estimation and variable selection in state-space models for neural interfaces. IEEE Trans Biomed Eng. 2015 Feb;62(2):570-81. doi: 10.1109/TBME.2014.2360393. Epub 2014 Sep 26. PMID 25265627
- [Background] Pandarinath C, Gilja V, Blabe CH, Nuyujukian P, Sarma AA, Sorice BL, Eskandar EN, Hochberg LR, Henderson JM, Shenoy KV. Neural population dynamics in human motor cortex during movements in people with ALS. Elife. 2015 Jun 23;4:e07436. doi: 10.7554/eLife.07436. PMID 26099302
- [Background] Pandarinath C, O'Shea DJ, Collins J, Jozefowicz R, Stavisky SD, Kao JC, Trautmann EM, Kaufman MT, Ryu SI, Hochberg LR, Henderson JM, Shenoy KV, Abbott LF, Sussillo D. Inferring single-trial neural population dynamics using sequential auto-encoders. Nat Methods. 2018 Oct;15(10):805-815. doi: 10.1038/s41592-018-0109-9. Epub 2018 Sep 17. PMID 30224673
- [Background] Willett FR, Murphy BA, Young DR, Memberg WD, Blabe CH, Pandarinath C, Franco B, Saab J, Walter BL, Sweet JA, Miller JP, Henderson JM, Shenoy KV, Simeral JD, Jarosiewicz B, Hochberg LR, Kirsch RF, Ajiboye AB. A Comparison of Intention Estimation Methods for Decoder Calibration in Intracortical Brain-Computer Interfaces. IEEE Trans Biomed Eng. 2018 Sep;65(9):2066-2078. doi: 10.1109/TBME.2017.2783358. Epub 2017 Dec 14. PMID 29989927
- [Background] Brandman DM, Burkhart MC, Kelemen J, Franco B, Harrison MT, Hochberg LR. Robust Closed-Loop Control of a Cursor in a Person with Tetraplegia using Gaussian Process Regression. Neural Comput. 2018 Nov;30(11):2986-3008. doi: 10.1162/neco_a_01129. Epub 2018 Sep 14. PMID 30216140
- [Background] Vargas-Irwin CE, Feldman JM, King B, Simeral JD, Sorice BL, Oakley EM, Cash SS, Eskandar EN, Friehs GM, Hochberg LR, Donoghue JP. Watch, Imagine, Attempt: Motor Cortex Single-Unit Activity Reveals Context-Dependent Movement Encoding in Humans With Tetraplegia. Front Hum Neurosci. 2018 Nov 15;12:450. doi: 10.3389/fnhum.2018.00450. eCollection 2018. PMID 30524258
- [Background] Willett FR, Avansino DT, Hochberg LR, Henderson JM, Shenoy KV. High-performance brain-to-text communication via handwriting. Nature. 2021 May;593(7858):249-254. doi: 10.1038/s41586-021-03506-2. Epub 2021 May 12. PMID 33981047
- [Background] Deo DR, Rezaii P, Hochberg LR, M Okamura A, Shenoy KV, Henderson JM. Effects of Peripheral Haptic Feedback on Intracortical Brain-Computer Interface Control and Associated Sensory Responses in Motor Cortex. IEEE Trans Haptics. 2021 Oct-Dec;14(4):762-775. doi: 10.1109/TOH.2021.3072615. Epub 2021 Dec 17. PMID 33844633
- [Background] Simeral JD, Hosman T, Saab J, Flesher SN, Vilela M, Franco B, Kelemen JN, Brandman DM, Ciancibello JG, Rezaii PG, Eskandar EN, Rosler DM, Shenoy KV, Henderson JM, Nurmikko AV, Hochberg LR. Home Use of a Percutaneous Wireless Intracortical Brain-Computer Interface by Individuals With Tetraplegia. IEEE Trans Biomed Eng. 2021 Jul;68(7):2313-2325. doi: 10.1109/TBME.2021.3069119. Epub 2021 Jun 17. PMID 33784612
- [Background] Rastogi A, Willett FR, Abreu J, Crowder DC, Murphy BA, Memberg WD, Vargas-Irwin CE, Miller JP, Sweet J, Walter BL, Rezaii PG, Stavisky SD, Hochberg LR, Shenoy KV, Henderson JM, Kirsch RF, Ajiboye AB. The Neural Representation of Force across Grasp Types in Motor Cortex of Humans with Tetraplegia. eNeuro. 2021 Feb 19;8(1):ENEURO.0231-20.2020. doi: 10.1523/ENEURO.0231-20.2020. Print 2021 Jan-Feb. PMID 33495242
- [Background] Hosman T, Hynes JB, Saab J, Wilcoxen KG, Buchbinder BR, Schmansky N, Cash SS, Eskandar EN, Simeral JD, Franco B, Kelemen J, Vargas-Irwin CE, Hochberg LR. Auditory cues reveal intended movement information in middle frontal gyrus neuronal ensemble activity of a person with tetraplegia. Sci Rep. 2021 Jan 11;11(1):98. doi: 10.1038/s41598-020-77616-8. PMID 33431994
- [Background] Wilson GH, Stavisky SD, Willett FR, Avansino DT, Kelemen JN, Hochberg LR, Henderson JM, Druckmann S, Shenoy KV. Decoding spoken English from intracortical electrode arrays in dorsal precentral gyrus. J Neural Eng. 2020 Nov 25;17(6):066007. doi: 10.1088/1741-2552/abbfef. PMID 33236720
- [Background] Eichenlaub JB, Jarosiewicz B, Saab J, Franco B, Kelemen J, Halgren E, Hochberg LR, Cash SS. Replay of Learned Neural Firing Sequences during Rest in Human Motor Cortex. Cell Rep. 2020 May 5;31(5):107581. doi: 10.1016/j.celrep.2020.107581. PMID 32375031
- [Background] Stavisky SD, Willett FR, Avansino DT, Hochberg LR, Shenoy KV, Henderson JM. Speech-related dorsal motor cortex activity does not interfere with iBCI cursor control. J Neural Eng. 2020 Feb 5;17(1):016049. doi: 10.1088/1741-2552/ab5b72. PMID 32023225
- [Background] Rastogi A, Vargas-Irwin CE, Willett FR, Abreu J, Crowder DC, Murphy BA, Memberg WD, Miller JP, Sweet JA, Walter BL, Cash SS, Rezaii PG, Franco B, Saab J, Stavisky SD, Shenoy KV, Henderson JM, Hochberg LR, Kirsch RF, Ajiboye AB. Neural Representation of Observed, Imagined, and Attempted Grasping Force in Motor Cortex of Individuals with Chronic Tetraplegia. Sci Rep. 2020 Jan 29;10(1):1429. doi: 10.1038/s41598-020-58097-1. PMID 31996696
- [Background] Stavisky SD, Willett FR, Wilson GH, Murphy BA, Rezaii P, Avansino DT, Memberg WD, Miller JP, Kirsch RF, Hochberg LR, Ajiboye AB, Druckmann S, Shenoy KV, Henderson JM. Neural ensemble dynamics in dorsal motor cortex during speech in people with paralysis. Elife. 2019 Dec 10;8:e46015. doi: 10.7554/eLife.46015. PMID 31820736
- [Background] Willett FR, Young DR, Murphy BA, Memberg WD, Blabe CH, Pandarinath C, Stavisky SD, Rezaii P, Saab J, Walter BL, Sweet JA, Miller JP, Henderson JM, Shenoy KV, Simeral JD, Jarosiewicz B, Hochberg LR, Kirsch RF, Bolu Ajiboye A. Principled BCI Decoder Design and Parameter Selection Using a Feedback Control Model. Sci Rep. 2019 Jun 20;9(1):8881. doi: 10.1038/s41598-019-44166-7. PMID 31222030
- [Background] Milekovic T, Bacher D, Sarma AA, Simeral JD, Saab J, Pandarinath C, Yvert B, Sorice BL, Blabe C, Oakley EM, Tringale KR, Eskandar E, Cash SS, Shenoy KV, Henderson JM, Hochberg LR, Donoghue JP. Volitional control of single-electrode high gamma local field potentials by people with paralysis. J Neurophysiol. 2019 Apr 1;121(4):1428-1450. doi: 10.1152/jn.00131.2018. Epub 2019 Feb 20. PMID 30785814
- [Background] Young D, Willett F, Memberg WD, Murphy B, Rezaii P, Walter B, Sweet J, Miller J, Shenoy KV, Hochberg LR, Kirsch RF, Ajiboye AB. Closed-loop cortical control of virtual reach and posture using Cartesian and joint velocity commands. J Neural Eng. 2019 Apr;16(2):026011. doi: 10.1088/1741-2552/aaf606. Epub 2018 Dec 4. PMID 30523839
- [Background] Nuyujukian P, Albites Sanabria J, Saab J, Pandarinath C, Jarosiewicz B, Blabe CH, Franco B, Mernoff ST, Eskandar EN, Simeral JD, Hochberg LR, Shenoy KV, Henderson JM. Cortical control of a tablet computer by people with paralysis. PLoS One. 2018 Nov 21;13(11):e0204566. doi: 10.1371/journal.pone.0204566. eCollection 2018. PMID 30462658
- [Background] Rubin DB, Hosman T, Kelemen JN, Kapitonava A, Willett FR, Coughlin BF, Halgren E, Kimchi EY, Williams ZM, Simeral JD, Hochberg LR, Cash SS. Learned Motor Patterns Are Replayed in Human Motor Cortex during Sleep. J Neurosci. 2022 Jun 22;42(25):5007-5020. doi: 10.1523/JNEUROSCI.2074-21.2022. Epub 2022 May 19. PMID 35589391
- [Result] Simeral JD, Kim SP, Black MJ, Donoghue JP, Hochberg LR. Neural control of cursor trajectory and click by a human with tetraplegia 1000 days after implant of an intracortical microelectrode array. J Neural Eng. 2011 Apr;8(2):025027. doi: 10.1088/1741-2560/8/2/025027. Epub 2011 Mar 24. PMID 21436513
- [Result] Hochberg LR, Bacher D, Jarosiewicz B, Masse NY, Simeral JD, Vogel J, Haddadin S, Liu J, Cash SS, van der Smagt P, Donoghue JP. Reach and grasp by people with tetraplegia using a neurally controlled robotic arm. Nature. 2012 May 16;485(7398):372-5. doi: 10.1038/nature11076. PMID 22596161
- [Result] Jarosiewicz B, Masse NY, Bacher D, Cash SS, Eskandar E, Friehs G, Donoghue JP, Hochberg LR. Advantages of closed-loop calibration in intracortical brain-computer interfaces for people with tetraplegia. J Neural Eng. 2013 Aug;10(4):046012. doi: 10.1088/1741-2560/10/4/046012. Epub 2013 Jul 10. PMID 23838067
- [Result] Bacher D, Jarosiewicz B, Masse NY, Stavisky SD, Simeral JD, Newell K, Oakley EM, Cash SS, Friehs G, Hochberg LR. Neural Point-and-Click Communication by a Person With Incomplete Locked-In Syndrome. Neurorehabil Neural Repair. 2015 Jun;29(5):462-71. doi: 10.1177/1545968314554624. Epub 2014 Nov 10. PMID 25385765
- [Result] Gilja V, Pandarinath C, Blabe CH, Nuyujukian P, Simeral JD, Sarma AA, Sorice BL, Perge JA, Jarosiewicz B, Hochberg LR, Shenoy KV, Henderson JM. Clinical translation of a high-performance neural prosthesis. Nat Med. 2015 Oct;21(10):1142-5. doi: 10.1038/nm.3953. Epub 2015 Sep 28. PMID 26413781
- [Result] Ajiboye AB, Willett FR, Young DR, Memberg WD, Murphy BA, Miller JP, Walter BL, Sweet JA, Hoyen HA, Keith MW, Peckham PH, Simeral JD, Donoghue JP, Hochberg LR, Kirsch RF. Restoration of reaching and grasping movements through brain-controlled muscle stimulation in a person with tetraplegia: a proof-of-concept demonstration. Lancet. 2017 May 6;389(10081):1821-1830. doi: 10.1016/S0140-6736(17)30601-3. Epub 2017 Mar 28. PMID 28363483
- [Result] Pandarinath C, Nuyujukian P, Blabe CH, Sorice BL, Saab J, Willett FR, Hochberg LR, Shenoy KV, Henderson JM. High performance communication by people with paralysis using an intracortical brain-computer interface. Elife. 2017 Feb 21;6:e18554. doi: 10.7554/eLife.18554. PMID 28220753
- [Result] Brandman DM, Hosman T, Saab J, Burkhart MC, Shanahan BE, Ciancibello JG, Sarma AA, Milstein DJ, Vargas-Irwin CE, Franco B, Kelemen J, Blabe C, Murphy BA, Young DR, Willett FR, Pandarinath C, Stavisky SD, Kirsch RF, Walter BL, Bolu Ajiboye A, Cash SS, Eskandar EN, Miller JP, Sweet JA, Shenoy KV, Henderson JM, Jarosiewicz B, Harrison MT, Simeral JD, Hochberg LR. Rapid calibration of an intracortical brain-computer interface for people with tetraplegia. J Neural Eng. 2018 Apr;15(2):026007. doi: 10.1088/1741-2552/aa9ee7. PMID 29363625
- [Result] Rubin DB, Ajiboye AB, Barefoot L, Bowker M, Cash SS, Chen D, Donoghue JP, Eskandar EN, Friehs G, Grant C, Henderson JM, Kirsch RF, Marujo R, Masood M, Mernoff ST, Miller JP, Mukand JA, Penn RD, Shefner J, Shenoy KV, Simeral JD, Sweet JA, Walter BL, Williams ZM, Hochberg LR. Interim Safety Profile From the Feasibility Study of the BrainGate Neural Interface System. Neurology. 2023 Mar 14;100(11):e1177-e1192. doi: 10.1212/WNL.0000000000201707. Epub 2023 Jan 13. PMID 36639237
- [Derived] Singer-Clark T, Hou X, Card NS, Wairagkar M, Iacobacci C, Peracha H, Hochberg LR, Stavisky SD, Brandman DM. Speech motor cortex enables BCI cursor control and click. J Neural Eng. 2025 May 14;22(3):036015. doi: 10.1088/1741-2552/add0e5. PMID 40280150
- [Derived] Card NS, Wairagkar M, Iacobacci C, Hou X, Singer-Clark T, Willett FR, Kunz EM, Fan C, Vahdati Nia M, Deo DR, Srinivasan A, Choi EY, Glasser MF, Hochberg LR, Henderson JM, Shahlaie K, Stavisky SD, Brandman DM. An Accurate and Rapidly Calibrating Speech Neuroprosthesis. N Engl J Med. 2024 Aug 15;391(7):609-618. doi: 10.1056/NEJMoa2314132. PMID 39141853
- [Derived] Ali YH, Bodkin K, Rigotti-Thompson M, Patel K, Card NS, Bhaduri B, Nason-Tomaszewski SR, Mifsud DM, Hou X, Nicolas C, Allcroft S, Hochberg LR, Au Yong N, Stavisky SD, Miller LE, Brandman DM, Pandarinath C. BRAND: a platform for closed-loop experiments with deep network models. J Neural Eng. 2024 Apr 17;21(2):026046. doi: 10.1088/1741-2552/ad3b3a. PMID 38579696
- [Derived] Brandman DM, Cash SS, Hochberg LR. Review: Human Intracortical Recording and Neural Decoding for Brain-Computer Interfaces. IEEE Trans Neural Syst Rehabil Eng. 2017 Oct;25(10):1687-1696. doi: 10.1109/TNSRE.2017.2677443. Epub 2017 Mar 2. PMID 28278476
- [Derived] Willett FR, Pandarinath C, Jarosiewicz B, Murphy BA, Memberg WD, Blabe CH, Saab J, Walter BL, Sweet JA, Miller JP, Henderson JM, Shenoy KV, Simeral JD, Hochberg LR, Kirsch RF, Ajiboye AB. Feedback control policies employed by people using intracortical brain-computer interfaces. J Neural Eng. 2017 Feb;14(1):016001. doi: 10.1088/1741-2560/14/1/016001. Epub 2016 Nov 30. PMID 27900953
- See also: Home Page for BrainGate Research — http://www.braingate.org